CLINICAL TRIAL: NCT03449264
Title: Development of a Monocentric and Prospective Clinical and Biological Database in Digestive Cancers, Gynecological Cancers, Breast Cancers and Sarcomas
Brief Title: Development of Clinical and Biological Database
Acronym: BCBInstitut
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-URC2017/37
Record Dates: First submitted 2017-08-29; First posted 2018-02-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Digestive Cancer; Gynecologic Cancer; Breast Cancer; Sarcoma
MeSH Terms: conditions — Gastrointestinal Neoplasms; Breast Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): samples of different natures:
  * Tissue samples (tumor tissue and healthy tissue) frozen and secured in paraffin collected during surgery.
  * Blood samples taken at different times. During the blood samples taken for diagnosis and / or treatment, additional samples for research purposes will be carried out.
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Biological: biological collection

INTERVENTIONS:
Biological: biological collection — * Tissue samples (tumor tissue and healthy tissue) frozen and secured in paraffin collected during surgery.
  * Blood samples taken at different times. During the blood samples taken for diagnosis and / or treatment, additional samples for research purposes will be carried out.

SUMMARY:
The BCB is a tool:

* for research in analytical and public health epidemiology, biological research and for the development of data useful for clinical research and therapeutic trials;
* to help scientists understand and explain phenomena ranging from the interaction of molecules to the whole metabolism of the organism in normal and pathological situations;
* to identify potential strategies for prevention, diagnosis, management and analysis of cancer subtypes.

The creation of a broad clinical and biological prospective base dedicated to different types of cancer is essential for the development of such projects.

DETAILED DESCRIPTION:
Implementation of a translational research project is part of the Cancer Plan 2014-2019 and its axis 5 "Advancing clinical and translational research in oncology", and more precisely Action 5.1.

The national health strategy launched by the Minister of Health and the Minister of Research will allow a better integration between research, innovation, medicine and care for the benefit of patients and society.

Moreover, knowledge of mechanisms involved in the phenomena of tumor invasion, metastatic dissemination, resistance to treatment and companion testing is crucial for the emergence of new biomarkers and therapeutic innovation.

However, the study of the earliest phases of tumorigenesis as well as of the advanced stages of the disease are currently limited by the low availability of blood and tissue samples combined with quality and reliable clinical data.

To meet these demands, the research must then integrate databases creation open to researchers and the ongoing evaluation of the impact of projects on the health of cancer patients.

Integrated research associated with quality biological research is the guarantee of medical progress.

The multidisciplinary structure around collections of biological resources will enable the various actors to harmonize not only the collection but also the sharing of their data with a view to making them available for medico-scientific projects at a regional and national dimension. The Clinical Biological Database (BCB) should be used to identify and characterize new molecular markers for better diagnosis and / or treatment. It should also permit to optimize the collection of all this information, their integration and their transversal exploitation by different research disciplines (epidemiological, fundamental, translational, clinical).

The BCB is a tool:

* for research in analytical and public health epidemiology, biological research and for the development of data useful for clinical research and therapeutic trials;
* to help scientists understand and explain phenomena ranging from the interaction of molecules to the whole metabolism of the organism in normal and pathological situations;
* to identify potential strategies for prevention, diagnosis, management and analysis of cancer subtypes.

The creation of a broad clinical and biological prospective base dedicated to different types of cancer is essential for the development of such projects

ELIGIBILITY:
Inclusion Criteria:

* Age> at 18 years old,
* Patient with invasive or in situ tumor pathology (proven or suspected) any stage confounded,
* Patient in ICM at diagnosis

  * a digestive cancer (esophagus, stomach, pancreas, colon, rectum, anal canal) or
  * gynecological cancer (ovary, endometrium, cervix) or
  * breast cancer or
  * sarcoma.
* Naïve patient of any treatment for the present cancer,
* Patient requiring treatment involving at least one (or more) tumor surgery (s)
* Patient who has accepted supplementary blood samples,
* Patient having given his informed, written and express consent.

Exclusion Criteria:

* Patient not affiliated to a social protection scheme,
* Patient whose regular follow-up is a priori impossible for psychological, familial, social or geographical reasons,
* Pregnant and / or nursing women,
* Subject under tutelage, curatorship or safeguard of justice,
* Patient in an emergency situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2037-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who consent to participate in the study | through study completion, an average of 1 year
  the proportion of patients who consent to participate in the study among the screened patients

OTHER OUTCOMES:
Quality of life assessment at baseline for all participants in the study | through study completion, an average of 1 year
  Questionnaire assessment to measure the quality of life at baseline

CONTACTS AND LOCATIONS:
Overall Officials: jean pierre Bleuse, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut regional du Cancer - Val d Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No